CLINICAL TRIAL: NCT01120587
Title: The Start of Pharyngeal Phase of Swallowing in Healthy Individuals
Brief Title: Videofluoroscopic of Deglutition Study of the Initiation of Pharyngeal Phase in Young Adults
Acronym: VFD-IPP
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Izabella Santos Nogueira de Andrade, University of Fortaleza
Other Study IDs: 193/2006
Record Dates: First submitted 2010-05-10; First posted 2010-05-11 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-01

CONDITIONS: Young; Healthy
Keywords: Deglutition; Fluoroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study has as objective to characterize the start of pharyngeal phase of swallowing, in the various food consistencies and volumes, with and without the influence of verbal orders, observed on videofluoroscopy of deglutition.

DETAILED DESCRIPTION:
Quantitative study, transverse and observational study, in the period January to March 2010, in the Center Advanced Diagnosis and Treatment Trajan Almeida, in the city of Fortaleza, Ceará. The sample was composed by 40 individuals, with mean age 23.5 years, 35 (87.5 %) female and five (12.5%) male gender. was carried out an assessment videofluoroscopy swallowing in net consistencies (15 ml of water added to 15 ml of barium net), liquid paste (25ml of barium net), paste (two spoons of 5ml of thickening for 30ml of barium net) and solid (1/2 cracker waffer immersed the barium net), where the individuals remained seated and the images were carried out in the lateral position. From the beginning of the rapid movement of hyoid bone, verified the beginning of pharyngeal phase of swallowing in each consistency.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ages ranging between 20 and 30 years
* Without complaint of deglutition
* Not submitted to surgeries and/or other treatments in the region of head and neck, with the exception of dental equipment.

Exclusion Criteria:

* Individuals submitted to cardiac surgeries, chest and/or abdominal prior
* Patients with diabetes mellitus and/or neurological diseases beyond craniofacial abnormalities.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 Young adults and healthy, individuals with ages ranging between 20 and 30 years without, mean age 23.5 years, ranging between 20 and 30 years 87.5% (35/40) female 12.5% (5/40) male.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita de Cássia A Almeida, Graduate, Principal Investigator — Fortaleza University; Izabella SN Andrade, Master, Study Chair — University Fortaleza; Renata CB Haguette, Master, Study Chair — University Fortaleza